CLINICAL TRIAL: NCT05274126
Title: Implantation Sur Cinq Centres Médico-Psychologiques Franciliens du Parcours Socio-Sanitaire orienté Vers le Rétablissement (PASSVers2)
Brief Title: Implementation of a Social and Mental Health Support to Promote Recovery in Five Mental Health Facilities in Paris Area
Acronym: PASSVERS-2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Versailles Hospital (Other)
Collaborators: Agence régionale de santé Ile de France (Unknown); UNION NATIONALE DE FAMILLES ET AMIS DE PERSONNES MALADES ET/OU HANDICAPÉES PSYCHIQUES (Unknown)
Responsible Party: Principal Investigator, Dr Christine PASSERIEUX, Principal Investigator, Versailles Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: P20/03_ PASSVERS-2
Record Dates: First submitted 2022-02-15; First posted 2022-03-10 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Severe Mental Disorder
Keywords: Schizophrenia; Bipolar disorder; Autism
MeSH Terms: conditions — Mental Disorders; Schizophrenia; Bipolar Disorder; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: Prospective longitudinal uncontrolled multicenter study, with cohort follow-up, focusing on patients, professionals, relatives and structures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient group (single group) (Experimental): 300 Patients involved in the recovery process.
  Interventions: Behavioral: Patient group/Passvers

INTERVENTIONS:
Behavioral: Patient group/Passvers — Passvers intervention aims at :
  * helping patients followed in the centers, presenting a Severe and Persistent Mental Disorder (schizophrenia, mood disorder, autism spectrum disorder, etc.), at risk or in a situation of psychological disability, to enroll in a rehabilitation program towards recovery.
  * supporting the emergence and construction of projects by the people themselves, and to accompany them to realize them.
  * Encouraging the use of resources in their environment and common law mechanisms (city hall, department, associations, etc.) for better social integration.
  * encouraging involvement in care understood as useful tools for the realization of the personal project.
  Passvers also aims at :
  * promoting a change in professional practices within the team, in favor of recovery-oriented practices based on the concept of engagement or empowerment.
  * allowing cooperation between health and social structures aiming at destigmatizing mental illness.

SUMMARY:
Prospective longitudinal uncontrolled multicenter study, with cohort follow-up, focusing on patients, professionals, relatives and structures evolution during the implementation of recovery based intervention.

DETAILED DESCRIPTION:
This is a hybrid efficacy-implementation Type I recovery based interventional study based on a multicenter follow-up of a cohort of 300 patients with severe and persistent mental disorders (60 patients per center). The evolution of concepts and means of evaluation now allow a precise description of the mechanisms of recovery in all the diversity of its expression among patients, their entourages and the psychiatric facilities.

In the present study, the investigators aim to characterize simultaneously the patients' trajectories and the evolution of the care facilities and their professionals with respect to the principles of recovery. This double exploration should allow to build theoretical and practical references for the extension of this approach to other centers in France.

The study considers a dual timeline for data collection:

* The timeline associated with patients defined by the inclusion of each patient and extending to 24 months after, punctuated by an assessment at 12 months;
* The timeline of the inclusion centers and professionals involved in the rehabilitation projects defined by the beginning of the study and extending beyond the end of inclusion of the last patient, punctuated by annual intermediate evaluations of the means allocated by the structure and the positioning of the personnel in terms of recovery.

The intervention consists in a follow-up of the patients and their relatives by a psychiatric nurse and a social worker during 12 months. Both professionals, trained to rehabilitation and recovery principles, will focus on the patient's needs and goals in order to improve the outcome, quality-of-life and clinical status.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a severe and persistent mental disorder among the following ICD10 compliant diagnostic categories:

  * Schizophrenia spectrum disorder (F2x)
  * Recurrent or persistent mood disorders (F30.x, F31.x, F33.x, F34.x, F38.x)
  * Psychological developmental disorders including autism spectrum disorders (F8x) and childhood and adolescent onset disorders (F9x)
* Presence of an indication for inclusion in the rehabilitation project identified by the treating psychiatrist and endorsed in the inclusion session by the PASSVers staff.
* Written consent from the patient or his/her legal representative to participate in the study.

Exclusion Criteria:

* Presence of an not stabilized or progressive organic neurological pathology, neurodegenerative disease
* Psychological or behavioral disorders mainly related to addictions with substances
* Psychiatric disorders secondary to an organic pathology that is not stabilized or that is evolving
* The following psychiatric situations are reasons for non-inclusion in the absence of an argued and collegial reassessment (the reason being that, although PASSVers2 must be considered as a first intention proposal in many situations meeting the inclusion criteria, it cannot intervene or be thought of as a "solution" to certain complex situations):

  * Psychiatric disorders caused by pregnancy or immediate postpartum
  * Severe borderline personality disorder
  * Current suicidal crisis
  * Extreme fragility of the patient with respect to changes that may be induced by the project, associated with a high risk of self or hetero-aggression.
  * Patient under justice constraint
* Foreseeable departure from the geographic area, not allowing for certainty of further evaluation
* Refusal of the patient to be followed by a social-health team (i.e. refusal of care or refusal of a dialogue on social aspects and projects).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Patient self rating of recovery support by caregivers T0 | baseline
  5-item short version of INSPIRE measure (Brief INSPIRE), range from 5 to 25, 25 corresponds to maximal support
Patient self rating of recovery support by caregivers T12 | 1 year
  5-item short version of INSPIRE measure (Brief INSPIRE), range from 5 to 25, 25 corresponds to maximal support
Patient self rating of recovery support by caregivers and structure T0 | baseline
  Recovery Self-Assessment (RSA-R), range from 32 to 160, higher values correspond to more perceived help
Patient self rating of recovery support by caregivers and structure T12 | 1 year
  Recovery Self-Assessment (RSA-R), range from 32 to 160, higher values correspond to more perceived help
Patient functioning T0 | baseline
  Personal and Social Performance scale (PSP), range 0-100, 100 corresponds to better functioning
Patient functioning T12 | 1 year
  Personal and Social Performance scale (PSP), range 0-100, 100 corresponds to better functioning
Patient functioning T24 | 2 years
  Personal and Social Performance scale (PSP), range 0-100, 100 corresponds to better functioning
Patient self rating of quality of life T0 | baseline
  Shortened quality of life questionnaire (SQoL-18), range 18-90, higher values correspond to better quality of life
Patient self rating of quality of life T12 | 1 year
  Shortened quality of life questionnaire (SQoL-18), range 18-90, higher values correspond to better quality of life
Patient self rating of quality of life T24 | 2 years
  Shortened quality of life questionnaire (SQoL-18), range 18-90, higher values correspond to better quality of life
Psychotic symptoms T0 | baseline
  Positive and negative syndrome scale (PANSS), range 30-210, higher values correspond to higher symptoms levels
Psychotic symptoms T12 | 1 year
  Positive and negative syndrome scale (PANSS), range 30-210, higher values correspond to higher symptoms levels
Depression T0 | baseline
  Psychiatric symptoms scales rated by the clinicians (CDSS), range 0-27, higher values correspond to higher depressive symptoms
Depression T12 | 1 year
  Psychiatric symptoms scales rated by the clinicians (CDSS), range 0-27, higher values correspond to higher depressive symptoms
Clinical outcome T0: Clinically significant events | baseline
  Record of occurrences (boolean) and dates of any clinical event (hospitalizations, self-harming behavior) occurring during the course of the illness
Clinical outcome T12: Clinically significant events | 1 year
  Record of occurrences (boolean) and dates of any clinical event (hospitalizations, self-harming behavior) occurring during the course of the illness
Patient self rating of recovery T0 | baseline
  Questionnaire about the process of recovery (QPR), range from 22 to 110, higher values correspond to better recovery
Patient self rating of recovery T12 | 1 year
  Questionnaire about the process of recovery (QPR), range from 22 to 110, higher values correspond to better recovery
Patient self rating of recovery T24 | 2 years
  Questionnaire about the process of recovery (QPR), range from 22 to 110, higher values correspond to better recovery

SECONDARY OUTCOMES:
Professional's Recovery knowledge on patients T0 | baseline
  Recovery knowledge inventory (RKI), range 20-100, higher values correspond to better knowledge on recovery processes
Professional's Recovery knowledge on patients T12 | 1 year
  Recovery knowledge inventory (RKI), range 20-100, higher values correspond to better knowledge on recovery processes
Professional's Recovery opinions on patients T0 | baseline
  Practitioners' Beliefs, Goals and Practices in Psychiatric Rehabilitation (PBGP), range 26-104, higher values correspond to better views on patients recovery
Professional's Recovery opinions on patients T12 | 1 year
  Practitioners' Beliefs, Goals and Practices in Psychiatric Rehabilitation (PBGP), range 26-104, higher values correspond to better views on patients recovery
Stigmatization T0 | baseline
  Internalized stigma of mental illness: self-stigma (ISMI), range 29-116, higher values correspond to worse stigmatization perception
Stigmatization T12 | 1 year
  Internalized stigma of mental illness: self-stigma (ISMI), range 29-116, higher values correspond to worse stigmatization perception
Perceived needs T0 | baseline
  Perceived needs scale (ELADEB), Composite measure of perceived difficulty in meeting needs and needs of help
Perceived needs T12 | 1 year
  Perceived needs scale (ELADEB), Composite measure of perceived difficulty in meeting needs and needs of help
Goal achievement T12 | 1 year
  Goal achievement scale (GAS), range -2 to +2, higher values correspond to better achievement of one specific goal
Metacognitive strategies T0 | baseline
  Versailles Metacognitive Strategies Evaluation Questionnaire (V-MSEQ), range 25-175, higher values correspond to better metacognitive strategies
Sleep T0 | baseline
  Patient self rating of sleep (1 item Pittsburgh sleep quality index PSQI), range 1-4, lower values correspond to better sleep quality
Sleep T12 | 1 year
  Patient self rating of sleep (1 item Pittsburgh sleep quality index PSQI), range 1-4, lower values correspond to better sleep quality
Medication adherence T0 | baseline
  Medication Adherence Rating Scale (MARS), range 5-25, lower values correspond to better adherence to treatment
Medication adherence T12 | 1 year
  Medication Adherence Rating Scale (MARS), range 5-25, lower values correspond to better adherence to treatment
Illness severity T0 | baseline
  Clinical Global Impressions Scale (CGI-S), range 1-7, higher values correspond to more severe illness
Illness severity T12 | 1 year
  Clinical Global Impressions Scale (CGI-S), range 1-7, higher values correspond to more severe illness
Cognitive disability T0 | baseline
  Cognitive processes involved in disability in schizophrenia scale (CPSD), range 0-78, higher values correspond to better cognitive functioning
Cognitive disability T12 | 1 year
  Cognitive processes involved in disability in schizophrenia scale (CPSD), range 0-78, higher values correspond to better cognitive functioning
Entourage assessment of structure recovery orientation T0 | baseline
  Recovery Self-Assessment Significant other version (RSA-R entourage), range 40-200, higher values correspond to better recovery orientation
Entourage assessment of structure recovery orientation T12 | 1 year
  Recovery Self-Assessment Significant other version (RSA-R entourage), range 40-200, higher values correspond to better recovery orientation

OTHER OUTCOMES:
Structure recovery orientation T0 | baseline
  Recovery Self-Assessment Services (RSA-R Services), range 32-160, higher values correspond to more pronounced recovery orientation of the structure
Structure recovery orientation T24 | 2 years
  Recovery Self-Assessment Services (RSA-R Services), range 32-160, higher values correspond to more pronounced recovery orientation of the structure
Implementation fidelity T0 | baseline
  Professional ratings of Passvers fidelity scale, range 0-92, higher values correspond to better implementation
Implementation fidelity T24 | 2 years
  Professional ratings of Passvers fidelity scale, range 0-92, higher values correspond to better implementation

CONTACTS AND LOCATIONS:
Overall Officials: Christine Passerieux, Prof, Principal Investigator — CH Versailles
Locations (5):
- France (5):
  - Centre Hospitalier d'Argenteuil, secteurs 95G05, 95G06, 95G13,, Argenteuil
  - Hôpital Sainte Anne - GHU Paris Psychiatrie & Neurosciences, secteur G75015, Paris
  - Centre Hospitalier de Plaisir, secteur 78G16, CMP de Rambouillet, Rambouillet
  - Etablissement de Santé Mentale de Rueil-Malmaison, Groupe MGEN, secteur 92G13, CMP de Rueil-Malmaison, Rueil-Malmaison
  - Centre Hospitalier de Versailles, secteur 78G17, Centre Bleuler, Versailles, Versailles

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bazin, N. Les suivis sociosanitaires des personnes présentant un trouble mental sévère et persistant : expérimentation PASSVers à Versailles. Inf. Psychiatr. 95, 509-513 (2019).